CLINICAL TRIAL: NCT05067634
Title: Open-Label Safety and Efficacy Study of Cenobamate in Pediatric Subjects 2-17 Years of Age With Partial-onset (Focal) Seizures
Brief Title: Safety and Efficacy Study of Cenobamate in Pediatric Subjects 2-17 Years of Age With Partial-onset (Focal) Seizures
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YKP3089C040
Record Dates: First submitted 2021-09-14; First posted 2021-10-05 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Partial Epilepsy
Keywords: Partial-onset (focal) seizures; Pediatrics
MeSH Terms: conditions — Epilepsies, Partial; Seizures | interventions — Cenobamate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 12 to < 18 year olds (Experimental)
  Interventions: Drug: Xcopri
- 6 to <12 years old (Experimental)
  Interventions: Drug: Xcopri
- 4 to <6 years old (Experimental)
  Interventions: Drug: Xcopri
- 2 to <4 years old (Experimental)
  Interventions: Drug: Xcopri

INTERVENTIONS:
Drug: Xcopri — Age groups 12 to <18 will enroll once dosing data is received from Cohort I of the PK analysis of YKP3089C039 study. Age groups 6 to <12 will enroll once dosing data is received from Cohort IIa of the PK analysis of YKP3089C039 study. Age groups 4 to <6 will enroll once dosing data is received from Cohort IIb of the PK analysis of YKP3089C039 study. Age groups 2 to <4 will enroll once dosing data is received from Cohort III of the PK analysis of YKP3089C039 study.

SUMMARY:
Primary objective: To evaluate the safety and tolerability of cenobamate in pediatric subjects 2-17 years of age with partial-onset (focal) seizures

DETAILED DESCRIPTION:
Secondary objectives:

* To evaluate the efficacy of cenobamate tablets and suspension in pediatric subjects with partial onset (focal) seizures
* To evaluate the pharmacokinetics of cenobamate tablets and suspension in pediatric subjects with partial onset seizures
* To evaluate the PK/pharmacodynamics of cenobamate in pediatric subjects with partial onset (focal) seizures
* Acceptability and palatability assessment (determined by a 5-point Hedonic Scale) of the oral formulation and the 12.5 mg tablets - Day 1, and Day 15

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of epilepsy with partial-onset (focal) seizures (POS) with or without secondarily generalized seizures according to the International League Against Epilepsy's (ILAE) Classification of Epileptic Seizures. A diagnosis should have been established at least 12 months prior to Visit 1 (Screening) by clinical history and an electroencephalogram (EEG) that is consistent with the diagnosis; normal interictal EEGs will be allowed provided that the participant meets the other diagnosis criterion (i.e., clinical history)
2. Male or female participant, from age 2 to less than 18 years at the time of informed consent/assent (dates including informed consent in YKP3089C039)
3. Have a minimum weight of 10.0 kilograms (kg) (22.0 pounds [lb])
4. Have had a brain imaging (e.g., magnetic resonance imaging [MRI] scan or computed tomography (CT) within 10 years before Visit 1 (Screening) that ruled out a progressive cause of epilepsy.
5. For subjects new to Study YKP3089C040, participants must have had at least 1 POS seizure during the 28-day Baseline Period. Only simple POS with motor signs, complex POS, and complex POS with secondary generalization are counted toward this inclusion for POS
6. Are currently being treated with stable doses of 1 to a maximum of 3 approved antiepileptic drugs (AEDs). Doses must be stable for at least 4 weeks before to Visit 1 (Screening). A vagal nerve stimulator [VNS] will not be counted as one of the 3 allowed AEDs but the settings should be stable for at least 4 weeks prior to Visit 1 (Screening).
7. Investigator believes subject could benefit from new or continued exposure to study drug
8. Subjects entering from study YKP3089C039 must continue to meet all of the inclusion criteria from the YKP3089C039 study
9. Subjects receiving felbamate as a concomitant AED must meet the following criteria:

   1. Have a 12-month history of felbamate use and a history of a fixed dosing regimen for a minimum of 60 days prior to Visit 1 (Screening).
   2. No prior or known history of hepatotoxicity or hematologic disorder due to felbamate.
10. Subjects following a ketogenic diet will be allowed as long as the diet has been stable for at least 30 days prior to Visit 1 (Screening) and will remain stable for the duration of the study

Exclusion Criteria:

1. Females who are breastfeeding or pregnant at Screening or Baseline.
2. Current or history of pseudo-seizures (psychogenic nonepileptic seizures) within approximately 2 years before Visit 1 (Screening).
3. Have a history of status epilepticus that required hospitalization during the 6 months before Visit 1 (Screening).
4. Have an unstable psychiatric diagnosis that may confound participants' ability to participate in the study or that may prevent completion of the protocol-specified tests (e.g., significant suicide risk, including suicidal behavior and ideation within 6 months before Visit 1 (Screening), current psychotic disorder, acute mania).
5. Any suicidal ideation with intent, with or without a plan within 6 months before Visit 2 [i.e., answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the Columbia-Suicide Severity Rating Scale (C-SSRS) in participants aged 6 and above, if able].
6. Are scheduled and/or confirmed to have epilepsy surgery within 6 months after Visit 1 (Screening); however, those who have previously documented "failed" epilepsy surgery will be allowed.
7. Evidence of clinically significant disease (e.g., cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments.
8. Presence of only nonmotor simple partial seizures or primary generalized epilepsies.
9. Evidence of moderate or severe renal insufficiency as defined by estimated glomerular filtration rates (eGFRs) of 31 to < 60 "milliliters per minute (mL/min)" and < 30 mL/min, respectively.
10. Evidence of significant active hepatic disease. Stable elevation of liver enzymes, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) due to concomitant medication(s), will be allowed if they are less than 3 times the upper limit of normal (ULN).
11. Evidence of significant active hematological disease; white blood cell (WBC) count equal or less than 2500/µL (2.50 1E+09/liter [L]) or an absolute neutrophil count equal or less than 1000/µL (1.00 1E+09/L).
12. Subjects with Familial short QT syndrome.
13. Clinically significant electrocardiogram (ECG) abnormality, including prolonged corrected QT interval (QTc) defined as greater than 450 milliseconds (msec) or shortened corrected QT interval (QTc) defined as less than 340 msec.
14. Have a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors.
15. Subject has a history of any serious drug-induced hypersensitivity reaction (including, but not limited to, Stevens Johnson syndrome, toxic epidermal necrolysis, or DRESS) or any drug-related rash requiring hospitalization.
16. History of AED-associated rash that involved conjunctiva or mucosae.
17. History of more than one non-serious drug-related hypersensitivity reaction that required discontinuation of the medication.
18. Concomitant use of vigabatrin. Participants who took vigabatrin in the past must be off vigabatrin for at least 5 months before Visit 1 (Screening) and with documentation showing no evidence of a vigabatrin-associated clinically significant abnormality in a visual perimetry test.
19. A history of intermittent use of rescue benzodiazepines (i.e., 1 to 2 doses over a 24-hour period is considered a 1-time rescue) more than once within the 30 days prior to Visit 1(Screening).
20. A VNS implanted less than 5 months before Visit 1 (Screening) or changes in parameter less than 4 weeks before Visit 1 (or thereafter during the study).
21. History of or a concomitant medical condition that in the opinion of the investigator(s) would preclude the participant's participation in a clinical study or compromise the participant's ability to safely complete the study.
22. Have participated in a study involving administration of an investigational drug or device within 4 weeks before Visit 1 (Screening), or within approximately 5 half-lives of the previous investigational compound, whichever is longer.
23. Participants with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
24. For subjects new to Study YKP3089C040 previous exposure to cenobamate or sensitivity/allergy to components of the oral suspension.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events and SAEs | 3 Years
  Summary statistics for clinical laboratory test results and vital signs; and physical examination, neurologic examination and electrocardiogram (ECG) finding.of age with partial-onset (focal) seizures

SECONDARY OUTCOMES:
To collect plasma samples of cenobamate to support the evaluation of the pharmacokinetics of cenobamate tablets and suspension in pediatric subjects with partial onset (focal) seizures | 3 Years
  The area under the curve (AUC) of Xcopri after a single and multiple doses of Xcopri
Acceptability and palatability assessment (determined by a 5-point Hedonic Scale) of the oral formulation and tablets | 3 Years
  Testing to determine how patients respond to the taste and route of Xcopri

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kamin, MD, Study Director — SK Life Science, Inc.
Locations (55):
- United States (25):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - University of California Davis Health, Sacramento, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Augusta University Medical Center, Augusta, Georgia
  - Clinical Integrative Research Center of Atlanta, Sandy Springs, Georgia
  - Meridian Clinical Research - Savannah Neurology Specialists, Savannah, Georgia
  - Kentucky Clinic, Lexington, Kentucky
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Spectrum Health Hospitals Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of Missouri Health Care - Women's and Children's Hospital, Columbia, Missouri
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Northeast Regional Epilepsy Group - Morristown, Morristown, New Jersey
  - Boston Children's Health Physicians - Neurology at Hawthorne, Hawthorne, New York
  - Duke University Hospital, Durham, North Carolina
  - Akron Children's Hospital NeuroDevelopmental Science Center/Pediatric Neurology, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Child Neurology Consultants of Austin, Austin, Texas
  - Scottish Rite for Children, Dallas, Texas
  - MultiCare Institute - Mary Bridge Children's Neurology, Tacoma, Washington
- Australia (4):
  - Austin Health, Heidelberg
  - Royal Children's Hospital Melbourne, Parkville
  - Sydney Children's Hospital - Randwick, Randwick
  - Children's Health Queensland Hospital and Health Service, South Brisbane
- Germany (5):
  - Charite University Hospital, Berlin
  - Diakonie Kork, Kehl
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Neurologische Klinik und Poliklinik Interdisziplinäres Epilepsiezentrum München, Munich
  - Universitätsklinikum Tübingen, Tübingen
- Hungary (5):
  - Bethesda Gyermekkorhaz, Budapest
  - Országos Klinikai Idegtudományi Intézet, Neurológiai Osztály, Budapest
  - Semmelweis University Dept. Of Paediatrics, Budapest
  - Servus Salvus Egészségügyi Szolgáltató Kft., Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
- Poland (3):
  - Niepubliczny Zaklad Opieki Zdrowotnej - Centrum Neurologii Dzieciecej i Leczenia Padaczki, Kielce
  - Centrum Medyczne Plejady, Krakow
  - Wojewódzki Specjalistyczny Szpital Dziecięcy im. św. Ludwika w Krakowie, Krakow
- South Korea (6):
  - Chungbuk National University Hospital, Cheonju
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Spain (7):
  - Hospital Sant Joan de Déu Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - Instituto de Investigación Sanitaria de la Fundación Ramón Domínguez, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville